CLINICAL TRIAL: NCT02820051
Title: Non-anesthesiologist-administered Propofol is Not Related to a Higher Increase in Transcutaneous CO2 Pressure During the Flexible Bronchoscopy Compared to Guideline-based Sedation: A Randomized Controlled Trial
Brief Title: Non-anesthesiologist-administered Propofol During the Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Julio Edgardo González Aguirre, Dr., FCCP, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NM13-009
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Conscious Sedation Failure During Procedure
Keywords: bronchoscopy; conscious sedation; midazolam; patient comfort; propofol
MeSH Terms: interventions — Midazolam; Propofol; Nalbuphine; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): In the group of midazolam, the initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Intervention: Transcutaneous CO2 monitor
  Interventions: Device: Transcutaneous CO2 monitor; Drug: Midazolam; Drug: Nalbuphine; Drug: Lidocaine
- Propofol (Experimental): In the group of propofol, the starting dose was 0.1 mg /kg. Additional doses of 10 mg of propofol were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Intervention: Transcutaneous CO2 monitor
  Interventions: Device: Transcutaneous CO2 monitor; Drug: Propofol; Drug: Nalbuphine; Drug: Lidocaine

INTERVENTIONS:
Device: Transcutaneous CO2 monitor — Measurement and surveillance of transcutaneous CO2 pressure (PtcCO2) to determine PtcCO2 behavior for each sedation group.
  Other Names: SenTec digital monitoring and Stow-Severinghaus type sensor
Drug: Midazolam — The initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of three to four in the Observer´s assessment of alertness/ sedation scale.
  Other Names: Dormicum
  Arms: Midazolam
Drug: Propofol — The initial dose was 0.1 mg /kg. Additional doses of 10 mg of propofol were allowed to reach a score level of three to four in the Observer´s assessment of alertness/ sedation scale.
  Other Names: Diprivan
  Arms: Propofol
Drug: Nalbuphine — The starting dose was 2 mg with additional doses of 1 mg if it was necessary.
  Other Names: Nubain
Drug: Lidocaine — Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Other Names: Xylocaine

SUMMARY:
Flexible bronchoscopy (FB) is a fundamental procedure for the diagnosis and treatment of respiratory diseases. Although midazolam is the recommended sedative agent by most guidelines, propofol has gained popularity due a short recovery time, however, evidence to propofol use for sedation during FB is scarce. There is little evidence about transcutaneous CO2 pressure (PtcCO2) behavior among patients sedated with propofol when it is administered by non-anesthesiologist and in combination with intravenous opioids for analgesia and cough inhibition.

The investigators performed a randomized controlled trial to determine whether non-anesthesiology-administered balanced-sedation with propofol was related to high values of values of PtcCO2 compared with guideline-based sedation (midazolam and opioid). The investigators included data from outpatients 18 years or older with an indication for FB in a university hospital in northern of Mexico. Secondary outcomes were recuperation time, patient satisfaction and adverse effects.

DETAILED DESCRIPTION:
The investigators prospectively included ambulatory patients aged > 18 years with an indication for flexible bronchoscopy. Bronchoscopic procedures were performed by residents of Respiratory and Critical Care Medicine subspecialty under the supervision of an attendant professor in a university-tertiary-referral center in northern Mexico. Patients with tracheostomy, known allergy to drugs used during procedural sedation, inability to answer the satisfaction questionnaires, psychiatric illness, pregnancy, or with ASA class IV or V, were excluded.

Patients were randomly assigned to receive sedation with midazolam or propofol. In the group of midazolam the initial dose was 0.05 mg/kg and in propofol group, the starting dose was 0.1 mg /kg. Additional doses of the corresponding drug (2 mg of midazolam or 10 mg of propofol) were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Prior to insertion of the bronchoscope, lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nasal insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.

In both groups, transcutaneous CO2 measurement was carried out with the system SenTec digital monitoring (Artemis Medical, Kent, London) by applying a Stow-Severinghaus (V-Sign sensor) type sensor in the ear lobe. All patients received supplementary oxygen and were monitored with intermittent non-invasive blood pressure measurements every 3 min and with continuous EKG and SO2 surveillance.

The assessment of the state of residual sedation was performed with the Aldrete scale at five, 10 and 15 minutes after complete FB. At the time of discharge from the bronchoscopy suite, a satisfaction questionnaire was applied to patients.

Sedation and analgesia were prescribed by the resident responsible for conducting FB without the support of specialists in anesthesiology. One collaborator blinded to the study group to which each patient belonged recorded all data derived from the procedure. The Bronchoscopist was blinded to PtcCO2 values.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients aged > 18 years with an indication for flexible bronchoscopy.

Exclusion Criteria:

* tracheostomy
* known allergy to drugs used during procedural sedation
* inability to answer the satisfaction questionnaires
* psychiatric illness, pregnancy
* ASA class IV or V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Mercado, MD, Study Chair — UANL
Locations (1):
- UANL University Hospital, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercado-Longoria R, Armeaga-Azonos C, Tapia-Orozco J, Gonzalez-Aguirre JE. Non-anesthesiologist-administered Propofol is not Related to an Increase in Transcutaneous CO2 Pressure During Flexible Bronchoscopy Compared to Guideline-based Sedation: A Randomized Controlled Trial. Arch Bronconeumol. 2017 Sep;53(9):489-494. doi: 10.1016/j.arbres.2016.12.018. Epub 2017 Apr 12. English, Spanish. PMID 28410767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February and July 2014, we prospectively included ambulatory patients > 18 years of age with an indication for FB. Bronchoscopic procedures were performed by residents of Respiratory and Critical Care Medicine under the supervision of an attendant professor in a tertiary-referral university hospital in northern Mexico.
Groups:
- Midazolam: In the group of midazolam, the initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Intervention: Transcutaneous CO2 monitor
  Transcutaneous CO2 monitor: Measurement and surveillance of transcutaneous CO2 pressure (PtcCO2) to determine PtcCO2 behavior for each sedation group.
  Midazolam: The initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of three to four in the Observer´s assessment of alertness/ sedation scale
  Nalbuphine: The starting dose was 2 mg
- Propofol: In the group of propofol, the starting dose was 0.1 mg /kg. Additional doses of 10 mg of propofol were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Intervention: Transcutaneous CO2 monitor
  Transcutaneous CO2 monitor: Measurement and surveillance of transcutaneous CO2 pressure (PtcCO2) to determine PtcCO2 behavior for each sedation group.
  Propofol: The initial dose was 0.1 mg /kg. Additional doses of 10 mg of propofol were allowed to reach a score level of three to four in the Observer´s assessment of alertness/ sedation scale.
  Nalbuphine: The starting dose was 2 mg
Period: Overall Study
Arm/Group | Midazolam | Propofol
Started | 49 | 53
Completed | 42 | 49
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Population: We eliminated eleven patients due lost to follow-up due to sensor dysfunction (seven in the midazolam group and four in the propofol group); finally, we only analyze data from 91 patients (42 in Midazolam and 49 in Propofol groups, respectively).
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Propofol | Total
Number analyzed (Participants) | 42 | 49 | 91
Age, Categorical [Count of Participants; unit: Participants] — Population: Eleven patients were lost to follow-up due to sensor dysfunction (seven in the midazolam group and four in the propofol group)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 42 | 49 | 91
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Eleven patients were lost to follow-up due to sensor dysfunction (seven in the midazolam group and four in the propofol group)
  years | 51.1 (16) | 46.6 (16.3) | 48.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Eleven patients were lost to follow-up due to sensor dysfunction (seven in the midazolam group and four in the propofol group)
  Participants
    Female | 14 | 16 | 30
    Male | 28 | 33 | 61
Region of Enrollment [Number; unit: participants] — Population: Eleven patients were lost to follow-up due to sensor dysfunction (seven in the midazolam group and four in the propofol group)
  participants
    Mexico | 42 | 49 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change in Transcutaneous CO2 Pressure
Description: Our primary outcome was to assess the difference in PtCO2 values during and after FB between the groups. We hypothesized that PtcO2 values are not higher in patients who received NAAP balanced sedation.
Time Frame: Change from Baseline PtcCO2 (minute 0) to PtcCO2 at minute 60
Measure: Mean (Standard Deviation); unit: Unit of Measure "mmHg"
Arm/Group | Midazolam | Propofol
Number analyzed (Participants) | 42 | 49
Unit of Measure "mmHg" | 43.6 (7.5) | 45.6 (9.6)
Statistical Analysis 1: Comparison: Midazolam vs Propofol; The sample was calculated with alpha 0.05, beta 0.20, standard deviation of 7.3,8 minimum PtcCO2 difference to detect of 5 mmHg, loss to follow-up estimated 0.20, and two-tails. According to the above, the sample size was 42 patients per group; Test type: Superiority; p = 0.281, Wilcoxon (Mann-Whitney) — threshold for statistical significance: < 0.05; We tested normal distribution with the Kolmogorov-Smirnov test. Data are shown as means and standard deviations for variables with normal distribution and as medians and interquartile ranges for non-normal variables. We used the t-test, the Mann-Whitney U-test, ANOVA, or chi-square as indicated. We defined a statistically significant difference as a P value < 0.05. The analysis was performed using SPSS version 18.0 for Windows (SPSS Inc., Chicago, IL)

2. Secondary Outcome: Residual Sedation Assessed Using the Aldrete Scale
Description: The assessment of the state of residual sedation was performed with the Aldrete scale at minute 30 after complete bronchoscopy.
  The Aldrete's scoring system is a commonly used scale for determining when people can be safely discharged from the post-anesthesia care unit. The Minumum value is 0 points and the maximum value is 10 pots. Scores of 9 or greater allow patients to leave Post Anaesthetic Care Unit.
Time Frame: 30 min after ending of the bronchoscopy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Midazolam: In the group of midazolam, the initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of 3 to 4 in the Observer´s assessment of alertness/ sedation scale. All patients received nalbuphine in a starting dose of 2 mg with additional doses of 1 mg if it was necessary. Lidocaine spray was applied to the nasal mucosa and pharynx for bronchoscope nostril insertion, and only in the pharynx for bronchoscope oral insertion. Topical lidocaine was applied using the spray-as-you-go technique, at a maximum dose of 7 mg/kg.
  Intervention: Transcutaneous CO2 monitor
  Transcutaneous CO2 monitor: Measurement and surveillance of transcutaneous CO2 pressure (PtcCO2) to determine PtcCO2 behavior for each sedation group.
  Midazolam: The initial dose was 0.05 mg/kg. Additional doses of 2 mg of midazolam were allowed to reach a score level of three to four in the Observer´s assessment of alertness/ sedation scale.
  Nalbuphine: The starting dose was 2 mg
Arm/Group | Midazolam | Propofol
Number analyzed (Participants) | 42 | 49
score on a scale | 10 [9 to 10] | 10 [10 to 10]
Statistical Analysis 1: Comparison: Midazolam vs Propofol; Test type: Superiority — We used the t-test, the Mann-Whitney U-test, ANOVA, or chi-square as indicated. We defined a statistically significant difference as a P value < 0.05; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Patient Comfort Assessed Using a Satisfaction Questionnaire
Description: At the time of discharge from the bronchoscopy suite, satisfaction was assessed using a visual analog scale of 1 (not satisfied) to 10 (very satisfied).
Time Frame: at discharge from bronchoscopy suite, average 60 min from FB start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Midazolam | Propofol
Number analyzed (Participants) | 42 | 49
score on a scale | 8.41 (1.25) | 8.97 (0.98)
Statistical Analysis 1: Comparison: Midazolam vs Propofol; Test type: Superiority — T test; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During bronchoscopy study and at sedation recovery period (on average 60 minutes from the beginning of the procedure)
Arm/Group | Midazolam | Propofol
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/53
Other Adverse Events (participants affected / at risk) | 13/49 | 11/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=49) | Propofol (N=53)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
This study has several limitations: 1) it was not blinded, 2) All patients were ambulatory and with low or intermediate anesthetic risk. 3) In our bronchoscopy service, nalbuphine is the only opioid available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No